CLINICAL TRIAL: NCT05496504
Title: Incidence and Prognostic Significance of (Malignant) Arrhythmias During Repetitive Holter Electrocardiograms in Patients With Pulmonary Hypertension
Brief Title: Pulmonary Hypertension and Arrhythmia
Status: Completed | Type: Observational
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Collaborators: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: PH09_08_2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; PH; arrhythmias; survival
MeSH Terms: conditions — Hypertension, Pulmonary; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Holter ECG

SUMMARY:
Patients with pulmonary hypertension underwent (routine) Holter ECG and were screened for (malignant) arrhyhtmias. Results of Holter ECGs were correlated with clinicial and technical data (echocardiography and right heart catheterization).

ELIGIBILITY:
Inclusion Criteria: Holter ECG -

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PH of all groups
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Arrhythmias during Holter ECG | 1-3 day(s)
  Which kind of arrhythmias could be detected during repetitive Holter ECG in patients with PH?

SECONDARY OUTCOMES:
Relation between arrhythmias and PH group, echocardiographic data, right heart catheterization data. | 1-3 day(s)

IPD SHARING:
Plan to Share IPD: No